CLINICAL TRIAL: NCT04896008
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate Sotatercept When Added to Maximum Tolerated Background Therapy in Participants With Pulmonary Arterial Hypertension (PAH) World Health Organization (WHO) Functional Class (FC) III or FC IV at High Risk Mortality
Brief Title: A Study of Sotatercept in Participants With PAH WHO FC III or FC IV at High Risk of Mortality (MK-7962-006/ZENITH)
Acronym: ZENITH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Acceleron Pharma, Inc., a wholly-owned subsidiary of Merck & Co., Inc., Rahway, NJ USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 7962-006; A011-14 (Other: Acceleronpharma); MK-7962-006 (Other: MSD); 2023-509140-10-00 (Registry Identifier: EU CT); U1111-1309-6376 (Registry Identifier: UTN); 2021-001498-21 (EudraCT Number)
Record Dates: First submitted 2021-05-13; First posted 2021-05-21 (Actual); Results first posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Pulmonary, hypertension, sotatercept
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Hypertension | interventions — ACE-011

STUDY DESIGN:
Intervention Model Description: Each eligible participant will be randomized in a 1:1 ratio to 1 of the following 2 treatment arms during a double-blind placebo-controlled treatment period:
  * Sotatercept at a starting dose of 0.3 mg/kg, with a target dose of 0.7 mg/kg, subcutaneously (SC) every 21 days plus background PAH therapy; or
  * Placebo administered SC every 21 days plus background PAH therapy.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participants on background PAH therapy will be administered placebo by SC injection every 21 days
  Interventions: Other: Placebo
- Sotatercept (Experimental): Participants on background PAH therapy will be administered sotatercept by SC injection at a starting dose of 0.3 mg/kg, with a target dose of 0.7 mg/kg, every 21 days
  Interventions: Drug: Sotatercept

INTERVENTIONS:
Drug: Sotatercept — SC injection
  Other Names: MK-7962; ACE-011
  Arms: Sotatercept
Other: Placebo — Placebo-matched SC injection
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate the effects of sotatercept (MK-7962, formerly called ACE-011) treatment (plus maximum tolerated background pulmonary arterial hypertension [PAH] therapy) versus placebo (plus maximum tolerated background PAH therapy) on time to first event of all cause death, lung transplantation, or PAH worsening-related hospitalization of ≥24 hours, in participants with World Health Organization (WHO) functional class (FC) III or FC IV PAH at high risk of mortality.

DETAILED DESCRIPTION:
This is a phase 3, randomized, double-blind, placebo-controlled study to evaluate sotatercept when added to maximum tolerated background PAH therapy on time to first event of all-cause death, lung transplantation, or PAH worsening related hospitalization of ≥24 hours, in participants with WHO FC III PAH or WHO FC IV PAH at high risk of mortality.

Participants with symptomatic PAH (WHO FC III or FC IV at high risk of mortality) who present with idiopathic or heritable PAH, PAH associated with connective tissue diseases (CTD), drug- or toxin-induced, post-shunt correction PAH, or PAH presenting at least 1 year following the correction of congenital heart defect. Participants must have a Registry to Evaluate Early and Long-Term PAH Disease Management (REVEAL) Lite 2.0 risk score of ≥9 and be on maximum tolerated combination background PAH therapy.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnostic right heart catheterization prior to screening confirming the diagnosis of WHO PAH Group 1 in any of the following subtypes:

  * Idiopathic PAH
  * Heritable PAH
  * Drug/toxin-induced PAH
  * PAH associated with CTD
  * PAH associated with simple, congenital systemic to pulmonary shunts at least 1 year following repair
* Symptomatic PAH classified as WHO FC III or IV
* REVEAL Lite 2.0 risk score of ≥9
* Right heart catheterization performed during screening (or within 2 weeks prior to screening, if done at the clinical study site) documenting a minimum PVR of ≥5 Wood units and a pulmonary capillary wedge pressure (PCWP) or left ventricular end-diastolic pressure (LVEDP) of ≤15 mmHg
* Clinically stable and on stable doses of maximum tolerated (per investigator's judgment) double or triple background PAH therapies for at least 30 days prior to screening
* Females of childbearing potential must:

  * Have 2 negative urine or serum pregnancy tests as verified by the investigator prior to starting study therapy; must agree to ongoing urine or serum pregnancy testing during the course of the study and until 8 weeks after the last dose of the study drug
  * If sexually active with a male partner, have used, and agree to use highly effective contraception without interruption per protocol; for at least 28 days prior to starting the investigational product, during the study (including dose interruptions), and for 16 weeks (112 days) after discontinuation of study treatment
  * Refrain from breastfeeding a child or donating blood, eggs, or ovum for the duration of the study and for at least 16 weeks (112 days) after the last dose of study treatment
* Male participants must:

  * Agree to use a condom, defined as a male latex condom or nonlatex condom NOT made out of natural (animal) membrane (e.g., polyurethane), during sexual contact with a pregnant female or a female of childbearing potential while participating in the study, during dose interruptions, and for at least 16 weeks (112 days) following investigational product discontinuation, even if he has undergone a successful vasectomy
  * Refrain from donating blood or sperm for the duration of the study and for 16 weeks (112 days) after the last dose of study treatment
* Ability to adhere to study visit schedule and understand and comply with all protocol requirements
* Ability to understand and provide written informed consent

Exclusion Criteria:

* Diagnosis of pulmonary hypertension (PH) WHO Groups 2, 3, 4, or 5
* Diagnosis of the following PAH Group 1 subtypes: human immunodeficiency virus-associated PAH and PAH associated with portal hypertension
* Diagnosis of pulmonary veno-occlusive diseases or pulmonary capillary hemangiomatosis or overt signs of capillary and/or venous involvement
* Hemoglobin at screening above gender-specific upper limit of normal (ULN), per local laboratory test
* Baseline platelet count <50,000/mm3 (<50.0 x 109/L) at screening
* Baseline systolic blood pressure <85 mmHg at screening
* Pregnant or breastfeeding women
* Serum alanine aminotransferase or aspartate aminotransferase levels or total bilirubin >3.0×ULN
* Currently enrolled in or have completed any other investigational product study within 30 days for small molecule drugs or within 5 half-lives for biologics prior to the date of signed informed consent
* Prior exposure to sotatercept or known allergic reaction to sotatercept, its excipients or luspatercept
* History of pneumonectomy
* Untreated more than mild obstructive sleep apnea
* History of known pericardial constriction
* History of restrictive or congestive cardiomyopathy
* Electrocardiogram (ECG) with Fridericia's corrected QT interval (QTcF) >500 ms during the screening period
* Personal or family history of long QT syndrome or sudden cardiac death
* Left ventricular ejection fraction <45% on historical echocardiogram within 1 year prior to the screening visit
* Any current or prior history of symptomatic coronary disease (prior myocardial infarction, percutaneous coronary intervention, coronary artery bypass graft surgery, or cardiac anginal chest pain) in the past 6 months prior to the screening visit
* Cerebrovascular accident within 3 months prior to the screening visit
* Significant (≥ 2+ regurgitation) mitral regurgitation or aortic regurgitation valvular disease
* Currently on dialysis or anticipated need for dialysis within the next 12 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-07-26 (Actual); Study Completion 2025-02-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (57):
- United States (26):
  - Arizona Pulmonary Specialists ( Site 1010), Phoenix, Arizona
  - David Geffen School of Medicine at UCLA ( Site 1068), Los Angeles, California
  - University of California Irvine ( Site 1086), Orange, California
  - University of California San Diego Medical Center ( Site 1002), San Diego, California
  - University of California San Francisco ( Site 1019), San Francisco, California
  - University of Colorado Hospital ( Site 1013), Aurora, Colorado
  - The George Washington University Medical Faculty Associates ( Site 1025), Washington D.C., District of Columbia
  - Mayo Clinic Jacksonville - PPDS ( Site 1045), Jacksonville, Florida
  - AdventHealth Medical Group Advanced Lung Disease ( Site 1058), Orlando, Florida
  - Northside Hospital ( Site 1073), Atlanta, Georgia
  - University Of Iowa Hospitals and Clinics ( Site 1050), Iowa City, Iowa
  - University of Kansas Medical Center ( Site 1020), Kansas City, Kansas
  - Tufts Medical Center - PPDS ( Site 1012), Boston, Massachusetts
  - Brigham and Women's Hospital ( Site 1014), Boston, Massachusetts
  - University of Michigan ( Site 1011), Ann Arbor, Michigan
  - Washington University School of Medicine ( Site 1022), St Louis, Missouri
  - University of Nebraska Medical Center ( Site 1053), Omaha, Nebraska
  - University of New Mexico Health Sciences Center ( Site 1048), Albuquerque, New Mexico
  - University of Rochester Medical Center - PPDS ( Site 1039), Rochester, New York
  - Duke University Medical Center ( Site 1026), Durham, North Carolina
  - University of Cincinnati Medical Center ( Site 1035), Cincinnati, Ohio
  - The Cleveland Clinic Foundation. ( Site 1065), Cleveland, Ohio
  - Medical University of South Carolina - PPDS ( Site 1003), Charleston, South Carolina
  - Statcare Pulmonary Consultants - Knoxville ( Site 1031), Knoxville, Tennessee
  - University Of Texas Southwestern Medical Center ( Site 1038), Dallas, Texas
  - Medical College of Wisconsin - Froedtert Hospital ( Site 1051), Milwaukee, Wisconsin
- Australia (2):
  - St Vincent's Hospital Sydney ( Site 1102), Darlinghurst, New South Wales
  - John Hunter Hospital ( Site 1101), New Lambton Heights, New South Wales
- Belgium (2):
  - Hôpital Erasme ( Site 1402), Anderlecht, Bruxelles-Capitale, Region de
  - UZ Leuven Campus Gasthuisberg ( Site 1401), Leuven, Vlaams-Brabant
- Canada (2):
  - Peter Lougheed Centre ( Site 2102), Calgary, Alberta
  - Jewish General Hospital ( Site 2103), Montreal, Quebec
- France (7):
  - Hôpitaux Universitaires de Strasbourg ( Site 1307), Strasbourg, Bas-Rhin
  - Centre Hospitalier Universitaire de Toulouse. ( Site 1315), Toulouse, Haute-Garonne
  - CHU de Nancy - Hôpital de Brabois Adultes ( Site 1308), Vandœuvre-lès-Nancy, Meurthe-et-Moselle
  - CHRU Lille ( Site 1306), Lille, Nord
  - Hôpital Louis Pradel ( Site 1317), Bron, Rhone
  - CHU Bicêtre ( Site 1304), Le Kremlin-Bicêtre, Val-de-Marne
  - CHU de Poitiers ( Site 1316), Poitiers, Vienne
- Germany (7):
  - Thoraxklinik-Heidelberg gGmbH ( Site 1509), Heidelberg, Baden-Wurttemberg
  - Krankenhaus Neuwittelsbach ( Site 1510), München, Bavaria
  - Universitaetsklinikum Giessen und Marburg GmbH ( Site 1512), Giessen, Hesse
  - Medizinische Hochschule Hannover ( Site 1505), Hanover, Lower Saxony
  - Uniklinik Köln ( Site 1511), Cologne, North Rhine-Westphalia
  - Universitätsklinikum des Saarlandes ( Site 1513), Homburg, Saarland
  - Universitätsklinikum Carl Gustav Carus an der TU Dresden. ( Site 1501), Dresden, Saxony
- Lady Davis Carmel Medical Center ( Site 1705), Haifa, Israel
- Italy (2):
  - Ospedale S. Giuseppe Multimedica ( Site 2403), Milan, Lombardy
  - La Sapienza-Università di Roma-Policlinico Umberto I ( Site 2402), Roma
- Mexico (3):
  - Instituto Nacional De Cardiologia Dr. Ignacio Chavez ( Site 2503), Mexico City, Mexico City
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez" ( Site 2504), Monterrey, Nuevo León
  - Unidad de Investigación Clínica en Medicina, S.C ( Site 2505), Monterrey, Nuevo León
- VU Medisch Centrum ( Site 2601), Amsterdam, North Holland, Netherlands
- Hospital Universitario 12 de Octubre ( Site 1603), Madrid, Spain
- United Kingdom (3):
  - Royal Papworth Hospital ( Site 1208), Cambridge, Cambridgeshire
  - Royal Brompton Hospital ( Site 1206), London, London, City of
  - Imperial College Healthcare NHS Trust ( Site 1203), London, London, City of

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Result] Humbert M, McLaughlin VV, Badesch DB, Ghofrani HA, Gibbs JSR, Gomberg-Maitland M, Preston IR, Souza R, Waxman AB, Moles VM, Savale L, Vizza CD, Rosenkranz S, Shi Y, Miller B, Mackenzie HS, Kim SS, Loureiro MJ, Patel MJ, Koglin J, Cornell AG, Hoeper MM; ZENITH Trial Investigators. Sotatercept in Patients with Pulmonary Arterial Hypertension at High Risk for Death. N Engl J Med. 2025 May 29;392(20):1987-2000. doi: 10.1056/NEJMoa2415160. Epub 2025 Mar 31. PMID 40167274
- See also: Merck Clinical Trial Information — https://www.merckclinicaltrials.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of 255 screened participants, 173 were randomized. One participant was randomized in error and did not receive study treatment. This participant was discontinued from the study and no data was collected. As pre-specified in the statistical analysis plan (SAP), this participant was excluded from all study analyses. Therefore, analyses are presented for 172 participants.
Pre-assignment Details: Protocol-specified final analysis of all outcome measures is reported here. At the time of the primary completion data cutoff, 108 participants were ongoing in the study for safety and survival follow-up. Per protocol, participants completing this study may have been eligible to enroll in an open-label, long-term follow-up study (MK-7962-004; NCT04796337).
Groups:
- Sotatercept: Participants on background pulmonary arterial hypertension (PAH) therapy were administered sotatercept by subcutaneous (SC) injection at a starting dose of 0.3 mg/kg, with a target dose of 0.7 mg/kg, every 21 days for up to approximately 26 months.
- Placebo: Participants on background PAH therapy were administered placebo by SC injection every 21 days for up to approximately 26 months.
Period: Overall Study
Arm/Group | Sotatercept | Placebo
Started | 86 | 86
Completed | 4 | 30
Not Completed | 82 | 56
Not completed — Ongoing | 70 | 38
Not completed — Adverse Event | 0 | 2
Not completed — Death | 5 | 10
Not completed — More Than 3 Dose Delays Required Per Dose Adjustment Guidelines | 1 | 0
Not completed — Fridericia's Corrected QT Interval Above 500 ms | 0 | 1
Not completed — Unwillingness Or Inability To Comply With Protocol | 1 | 0
Not completed — Withdrawal by Subject | 1 | 4
Not completed — Investigator Decision | 2 | 0
Not completed — Transitioned to Commercial Sotatercept | 2 | 1

BASELINE CHARACTERISTICS:
Population: Of the 173 participants randomized in the study, one participant was randomized in error to the placebo arm and then immediately discontinued. This participant did not receive study treatment, and no data was collected. As pre-specified in the SAP, this participant was excluded from all study analyses. 4 participants were randomized in violation of the protocol with a REVEAL score of <9.
Groups:
- Sotatercept: Participants on background PAH therapy were administered sotatercept by subcutaneous (SC) injection at a starting dose of 0.3 mg/kg, with a target dose of 0.7 mg/kg, every 21 days for up to approximately 26 months.
- Total: Total of all reporting groups
Arm/Group | Sotatercept | Placebo | Total
Number analyzed (Participants) | 86 | 86 | 172
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.3 (14.3) | 53.5 (14.3) | 54.4 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 71 | 132
  Male | 25 | 15 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 12 | 18
  Not Hispanic or Latino | 78 | 73 | 151
  Unknown or Not Reported | 2 | 1 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 4 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 4 | 9
  White | 73 | 76 | 149
  West Indian | 1 | 0 | 1
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 2 | 1 | 3
Registry to Evaluate Early and Long-Term PAH Disease Management (REVEAL) Lite 2.0 Score [Count of Participants; unit: Participants] — PAH participants had REVEAL scores based on 6 variables (sub-score ranges): estimated glomerular filtration rate (eGFR) (0, +1), WHO functional class (FC) (-1, 0, +1, +2), systolic blood pressure (SBP) (0, +1), heart rate (0, +1), 6-minute walk distance (6MWD) (-2, -1, 0, +1), and N-terminal prohormone B-type natriuretic peptide (NT-proBNP) (-2, 0, +2). All sub-scores are added to a base score of +6 and a total REVEAL score of 1 to 14 is obtained (≤5 = low risk; 6,7 = intermediate risk; ≥8 = high risk). 4 participants were randomized in violation of the protocol with a REVEAL score of <9.
  Participants
    <9 | 1 | 3 | 4
    9 to 10 | 59 | 57 | 116
    ≥11 | 26 | 26 | 52
PAH Subtype [Count of Participants; unit: Participants] — Participants who were eligible for this study presented with symptomatic PAH that was classified as idiopathic, heritable, drug- or toxin-induced, associated with connective tissue disease, or post-shunt correction.
  Participants
    Idiopathic PAH | 42 | 44 | 86
    Heritable PAH | 11 | 7 | 18
    Drug or toxin-induced PAH | 6 | 5 | 11
    PAH associated with connective tissue disease | 22 | 26 | 48
    PAH associated with simple, congenital systemic-to-pulmonary shunts >1 year following shunt repair | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Time to First Confirmed Morbidity or Mortality Event
Description: Morbidity or mortality events were defined as all-cause death, lung transplantation, or PAH worsening-related hospitalization of ≥24 hours. All events were adjudicated by a blinded, independent committee of clinical experts. Only adjudication-confirmed lung transplantation and PAH worsening-related hospitalization of ≥24 hours were included in the primary analysis. All deaths that are a first event for a participant were included regardless of adjudication. The time from randomization to the first confirmed morbidity or mortality event, calculated using the non-parametric Kaplan-Meier method, is presented.
Time Frame: Up to approximately 26 months
Population: All randomized participants who received at least one dose of study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sotatercept | Placebo
Number analyzed (Participants) | 86 | 86
Months | NA [NA to NA] — NA = Median, upper limit, and lower limit not reached at time of data cut-off due to insufficient number of participants with an event. | 9.6 [6.2 to 14.8]
Statistical Analysis 1: Comparison: Sotatercept vs Placebo; Test type: Superiority; p < 0.0001, Log Rank — One-sided p-value based on log-rank test stratified by the randomization stratification factors (REVEAL Lite 2.0 risk score and PAH subtype); Hazard Ratio (HR) = 0.24, 95% CI 2-sided [0.13 to 0.43] — HR and associated 95% confidence interval were based on Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by the randomization stratification factors (REVEAL Lite 2.0 risk score and PAH subtype)

2. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to death due to any cause. As pre-specified in the SAP, all deaths up to data cutoff, including among participants who completed or discontinued the study, were included except for those that occurred after enrollment in the long-term follow-up study (MK-7962-004) or after lung transplantation. The OS for participants, calculated using the non-parametric Kaplan-Meier method, is reported.
Time Frame: Up to approximately 26 months
Population: All randomized participants who received at least one dose of study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sotatercept | Placebo
Number analyzed (Participants) | 86 | 86
Months | NA [NA to NA] — NA = Median, upper limit, and lower limit not reached at time of data cut-off due to insufficient number of participants with an event. | NA [NA to NA] — NA = Median, upper limit, and lower limit not reached at time of data cut-off due to insufficient number of participants with an event.
Statistical Analysis 1: Comparison: Sotatercept vs Placebo; Test type: Superiority; p = 0.0313, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.42, 95% CI 2-sided [0.17 to 1.07] — Based on Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by the randomization stratification factors (REVEAL Lite 2.0 risk score and PAH subtype)

3. Secondary Outcome: Transplant-free Survival
Description: Transplant-free survival was defined as the time from randomization to the first lung transplantation or death due to any cause. As pre-specified in the SAP, all deaths up to data cutoff, including among participants who completed or discontinued the study, were included except for those that occurred after enrollment in the long-term follow-up study (MK-7962-004) or after lung transplantation. Transplant-free survival for participants, calculated using the non-parametric Kaplan-Meier method, is reported.
Time Frame: Up to approximately 26 months
Population: All randomized participants who received at least one dose of study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sotatercept | Placebo
Number analyzed (Participants) | 86 | 86
Months | NA [NA to NA] — NA = Median, upper limit, and lower limit not reached at time of data cut-off due to insufficient number of participants with an event. | NA [8.8 to NA] — NA = Median and upper limit not reached at time of data cut-off due to insufficient number of participants with an event.
Statistical Analysis 1: Comparison: Sotatercept vs Placebo; Test type: Superiority; p = 0.0039, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.34, 95% CI 2-sided [0.15 to 0.78] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Percentage of Participants Who Experienced a Mortality Event
Description: Mortality events were defined as death due to any cause throughout the study. As pre-specified in the SAP, all deaths up to data cutoff, including among participants who completed or discontinued the study, were included except for those that occurred after enrollment in the long-term follow-up study (MK-7962-004) or after lung transplantation. The percent of participants who experienced a mortality event is reported.
Time Frame: Up to approximately 26 months
Population: All randomized participants who received at least one dose of study treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Sotatercept | Placebo
Number analyzed (Participants) | 86 | 86
Percentage of Participants | 8.1 | 15.1
Statistical Analysis 1: Comparison: Sotatercept vs Placebo; Test type: Superiority; p = 0.135, Cochran-Mantel-Haenszel — Two-sided p-value is calculated based on Cochran-Mantel-Haenszel method stratified by the randomization stratification factors (REVEAL Lite 2.0 risk score and PAH subtype); Treatment Difference = -7.29, 95% CI 2-sided [-17.65 to 2.41] — Based on Miettinen and Nurminen method stratified by the randomization stratification factors (REVEAL Lite 2.0 risk score and PAH subtype)

5. Secondary Outcome: Change From Baseline in REVEAL Lite 2.0 Risk Score at Week 24
Description: REVEAL Lite 2.0 risk scoring is used to guide PAH treatment decisions. Total score uses 6 variables with each assessed based on contribution to mortality risk. Variables and sub-score ranges: eGFR (0, +1), WHO FC (-1, 0, +1, +2), SBP (0, +1), heart rate (0, +1), 6MWD (-2, -1, 0, +1), and NT-proBNP (-2, 0, +2). Sub-scores are added to a base score of +6 and a total score of 1 to 14 is obtained (≤5=low risk; 6,7=intermediate risk; ≥8=high risk). A higher score = higher risk. Per SAP, multiple imputation was used to impute the missing data at Week 24 for reasons other than death or a non-fatal clinical worsening event. Range was based on the minimum and maximum of median scores across the imputed dataset (100 repetitions). Thus, median change from baseline and range could be the same or show minimal variability. Comparisons with other REVEAL analyses may not be possible due to Week 24 data imputation. The change from baseline in REVEAL Lite 2.0 risk score at Week 24 is reported.
Time Frame: Baseline and Week 24
Population: All randomized participants who received at least one dose of study treatment and who were randomized more than 24 weeks prior to the data cutoff.
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | Sotatercept | Placebo
Number analyzed (Participants) | 77 | 78
Scores on a scale | -3.0 [-3.0 to -2.0] | 0.0 [0.0 to 0.0]
Statistical Analysis 1: Comparison: Sotatercept vs Placebo; Test type: Superiority; p < 0.001, Aligned Rank Stratified Wilcoxon — Two-sided p-value is provided using aligned rank stratified Wilcoxon test stratified by a randomization stratification factor (PAH subtype); Treatment Difference = -3.10, 95% CI 2-sided [-4.25 to -1.88] — Hodges-Lehmann location shift estimate with 95% CI is provided using aligned rank stratified Wilcoxon test stratified by a randomization stratification factor (PAH subtype)

6. Secondary Outcome: Percentage of Participants Achieving a Low or Intermediate (≤7) REVEAL Lite 2 Risk Score at Week 24
Description: REVEAL Lite 2.0 risk scoring is used to guide PAH treatment decisions. Total score uses 6 variables with each assessed based on contribution to mortality risk. Variables and sub-score ranges: eGFR (0, +1), WHO FC (-1, 0, +1, +2), SBP (0, +1), heart rate (0, +1), 6MWD (-2, -1, 0, +1), and NT-proBNP (-2, 0, +2). Sub-scores are added to a base score of +6 and a total score of 1 to 14 is obtained (≤5=low risk; 6,7=intermediate risk; ≥8=high risk). A higher score = higher risk. Per SAP, participants who did not have a REVEAL risk score at Week 24 were considered as non-responders and multiple imputation was not conducted for this endpoint. Comparisons between this analysis reporting non-imputed data should not be made to other REVEAL analyses which included imputation of missing Week 24 data. The percentage of participants who achieved a low or intermediate REVEAL Lite 2.0 score at Week 24 is reported.
Time Frame: Baseline and Week 24
Population: All randomized participants who received at least one dose of study treatment, who were randomized more than 24 weeks prior to the data cutoff, and who had a REVEAL Lite 2.0 risk score >7 at baseline.
Measure: Number; unit: Percentage of Participants
Arm/Group | Sotatercept | Placebo
Number analyzed (Participants) | 69 | 72
Percentage of Participants | 49.3 | 15.3
Statistical Analysis 1: Comparison: Sotatercept vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Two-sided p-value is calculated based on Cochran-Mantel-Haenszel method stratified by a randomization stratification factor (PAH subtype); Treatment Difference = 33.05, 95% CI 2-sided [18.41 to 46.98] — Based on Miettinen and Nurminen method stratified by a randomization stratification factors (PAH subtype)

7. Secondary Outcome: Change From Baseline in NT-proBNP Levels at Week 24
Description: NT-proBNP is secreted by cardiomyocytes in response to ventricular stretch and is an established noninvasive marker of ventricular dysfunction in patients with PAH. Blood samples were collected at baseline and at Week 24 to measure NT-proBNP levels. Per SAP, multiple imputation was used to impute the missing data at Week 24 for reasons other than death or a non-fatal clinical worsening event. Range was based on the minimum and maximum of median scores across the imputed dataset (100 repetitions). Thus, median change from baseline and range could be the same or show minimal variability. The change from baseline in NT-proBNP levels at Week 24 is reported.
Time Frame: Baseline and Week 24
Population: as for outcome 5
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Sotatercept | Placebo
Number analyzed (Participants) | 77 | 78
pg/mL | -1233.0 [-1233.0 to -1233.0] | 255.4 [211.0 to 263.0]
Statistical Analysis 1: Comparison: Sotatercept vs Placebo; Test type: Superiority; p < 0.001, Aligned Rank Stratified Wilcoxon — Two-sided p-value is provided using aligned rank stratified Wilcoxon test stratified by the randomization stratification factors (REVEAL Lite 2.0 risk score and PAH subtype); Treatment Difference = -2339.10, 95% CI 2-sided [-3378.74 to -1299.44] — Hodges-Lehmann location shift estimate with 95% CI is provided using aligned rank stratified Wilcoxon test stratified by the randomization stratification factors (REVEAL Lite 2.0 risk score and PAH subtype)

8. Secondary Outcome: Change From Baseline in Mean Pulmonary Artery Pressure (mPAP) at Week 24
Description: mPAP is a prognostic hemodynamic parameter measured at baseline and at Week 24 by right heart catheterization (RHC). Per SAP, multiple imputation was used to impute the missing data at Week 24 for reasons other than death or a non-fatal clinical worsening event. Range was based on the minimum and maximum of median scores across the imputed dataset (100 repetitions). Thus, median change from baseline and range could be the same or show minimal variability. The change from baseline in mPAP at Week 24 is reported.
Time Frame: Baseline and Week 24
Population: as for outcome 5
Measure: Median (Full Range); unit: mmHg
Arm/Group | Sotatercept | Placebo
Number analyzed (Participants) | 77 | 78
mmHg | -13.6 [-14.0 to -13.0] | 5.5 [5.0 to 6.0]
Statistical Analysis 1: Comparison: Sotatercept vs Placebo; Test type: Superiority; p < 0.001, Aligned Rank Stratified Wilcoxon — [p-value comment as in outcome 7, analysis 1]; Treatment Difference = -21.20, 95% CI 2-sided [-27.78 to -14.59] — [estimate comment as in outcome 7, analysis 1]

9. Secondary Outcome: Change From Baseline in Pulmonary Vascular Resistance (PVR)
Description: PVR is a prognostic hemodynamic variable of pulmonary circulation and was measured at baseline and at Week 24 by right heart catheterization (RHC). Per SAP, multiple imputation was used to impute the missing data at Week 24 for reasons other than death or a non-fatal clinical worsening event. Range was based on the minimum and maximum of median scores across the imputed dataset (100 repetitions). Thus, median change from baseline and range could be the same or show minimal variability. The change from baseline in PVR at Week 24 is reported.
Time Frame: Baseline and Week 24
Population: as for outcome 5
Measure: Median (Full Range); unit: Dynes*sec/cm^5
Arm/Group | Sotatercept | Placebo
Number analyzed (Participants) | 77 | 78
Dynes*sec/cm^5 | -156.6 [-160.0 to -152.0] | 46.6 [36.0 to 104.0]
Statistical Analysis 1: Comparison: Sotatercept vs Placebo; Test type: Superiority; p < 0.001, Aligned Rank Stratified Wilcoxon — [p-value comment as in outcome 7, analysis 1]; Treatment Difference = -339.60, 95% CI 2-sided [-511.09 to -168.06] — [estimate comment as in outcome 7, analysis 1]

10. Secondary Outcome: Percentage of Participants Who Improve in WHO FC
Description: The severity of a participant's PAH symptoms was graded using the WHO FC system. WHO functional classification for PAH ranges from Class I (no limitation in physical activity, no dyspnea with normal activity), Class II (slight limitation of physical activity), Class III (marked limitation of physical activity), and Class IV (cannot perform a physical activity without any symptoms, dyspnea at rest). Participants who improve in WHO FC were classified into "Improved", "No change", or "Worsened" (Improved = reduction in FC; Worsened = increase in FC; No change = no change in FC). The percentage of participants who had improvement from baseline in WHO FC at the end of the treatment period is reported.
Time Frame: Baseline and up to approximately 26 months
Population: All randomized participants who received at least one dose of study treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Sotatercept | Placebo
Number analyzed (Participants) | 86 | 86
Percentage of Participants | 55.8 | 27.9
Statistical Analysis 1: Comparison: Sotatercept vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 4, analysis 1]; Treatment Difference = 27.41, 95% CI 2-sided [12.85 to 40.98] — [estimate comment as in outcome 4, analysis 1]

11. Secondary Outcome: Change From Baseline in 6MWD at Week 24
Description: 6MWD was measured using the 6-Minute Walk Test (6MWT). The 6MWT measures the distance covered in 6 minutes and is intended to measure changes in functional exercise capacity. Each participant's 6MWD was measured at baseline and at 24 weeks. An increase in the distance walked during the 6MWT indicated improvement in functional exercise capacity. Per SAP, multiple imputation was used to impute the missing data at Week 24 for reasons other than death or a non-fatal clinical worsening event. Range was based on the minimum and maximum of median scores across the imputed dataset (100 repetitions). Thus, median change from baseline and range could be the same or show minimal variability. The change from baseline in 6MWD at Week 24 is reported.
Time Frame: Baseline and Week 24
Population: as for outcome 5
Measure: Median (Full Range); unit: Meters
Arm/Group | Sotatercept | Placebo
Number analyzed (Participants) | 77 | 78
Meters | 45.39 [45.00 to 46.00] | -5.36 [-9.50 to -1.00]
Statistical Analysis 1: Comparison: Sotatercept vs Placebo; Test type: Superiority; p < 0.001, Aligned Rank Stratified Wilcoxon — Two-sided p-value is provided using aligned rank stratified Wilcoxon test stratified by randomization stratification factor (REVEAL Lite 2.0 risk score and PAH subtype); Treatment Difference = 63.00, 95% CI 2-sided [23.22 to 102.73] — Hodges-Lehmann location shift estimate with 95% CI is provided using aligned rank stratified Wilcoxon test stratified by randomization stratification factor (REVEAL Lite 2.0 risk score and PAH subtype)

12. Secondary Outcome: Change From Baseline in Cardiac Output (CO) at Week 24
Description: CO is a prognostic hemodynamic parameter measured at baseline and at Week 24 by RHC. Per SAP, multiple imputation was used to impute the missing data at Week 24 for reasons other than death or a non-fatal clinical worsening event. Range was based on the minimum and maximum of median scores across the imputed dataset (100 repetitions). Thus, median change from baseline and range could be the same or show minimal variability. The change from baseline in CO at Week 24 is reported.
Time Frame: Baseline and Week 24
Population: as for outcome 5
Measure: Median (Full Range); unit: Liters/minute
Arm/Group | Sotatercept | Placebo
Number analyzed (Participants) | 77 | 78
Liters/minute | -0.1 [-0.1 to -0.1] | -0.38 [-0.42 to -0.35]
Statistical Analysis 1: Comparison: Sotatercept vs Placebo; Test type: Superiority; p = 0.119, Aligned Rank Stratified Wilcoxon — [p-value comment as in outcome 11, analysis 1]; Treatment Difference = 0.50, 95% CI 2-sided [-0.18 to 1.16] — [estimate comment as in outcome 11, analysis 1]

13. Secondary Outcome: Change From Baseline in European Quality of Life (EuroQoL)-5 Dimensions-5 Levels (EQ-5D-5L) Index Score at Week 24
Description: EQ-5D-5L is a standardized measure of health status, consisting of 5 health dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), each assessed on a 5-point scale (1=no problem, 2=slight problems, 3=moderate problems, 4=severe problems, 5=extreme problems). Participants score each dimension based on their health that day and their responses are used to generate a health index score. Index scores could range from <0 (a health state equivalent to dead with negative values representing a state worse than dead) to 1 (full health). Higher scores indicated better health and a positive change in score indicated improved overall health. Per SAP, multiple imputation was used to impute missing data at Week 24 for reasons other than death or a non-fatal clinical worsening event. Range was based on the minimum and maximum of median scores across the imputed dataset (100 repetitions). The change from baseline to Week 24 in EQ-5D-5L index score is reported.
Time Frame: Baseline and Week 24
Population: All randomized participants who received at least one dose of study treatment, who were randomized more than 24 weeks prior to the data cutoff, and who had data available from at least one baseline and post-baseline PRO assessment.
Measure: Median (Full Range); unit: Scores on a Scale
Arm/Group | Sotatercept | Placebo
Number analyzed (Participants) | 41 | 36
Scores on a Scale | 0.060 [-1.020 to 0.512] | 0.007 [-0.358 to 0.740]

ADVERSE EVENTS:
Time Frame: Up to approximately 27 months
Description: All-cause mortality was reported for all randomized participants. Serious AEs and Other AEs were reported for all randomized participants who received at least 1 dose of study treatment.
Arm/Group | Sotatercept | Placebo
All-Cause Mortality (participants affected / at risk) | 8/86 | 18/86
Serious Adverse Events (participants affected / at risk) | 46/86 | 55/86
Other Adverse Events (participants affected / at risk) | 79/86 | 74/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sotatercept (N=86) | Placebo (N=86)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 4 (4) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 2 (3)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 4 (4) | 9 (11)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (3)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 2 (2)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Right ventricular failure (Cardiac disorders) | 2 (2) | 11 (12)
Sinus node dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 3 (4) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 1 (3) | 0 (0)
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemoperitoneum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1)
Complication associated with device (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Sudden death (General disorders) | 0 (0) | 1 (1)
Vascular device occlusion (General disorders) | 1 (1) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis viral (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 2 (2) | 1 (1)
Diarrhoea infectious (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis norovirus (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Klebsiella bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2)
Perirectal abscess (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 7 (7) | 4 (4)
Pneumonia parainfluenzae viral (Infections and infestations) | 1 (1) | 0 (0)
Pseudomonas infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 3 (3) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 1 (1)
Spinal empyema (Infections and infestations) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0)
Vascular device infection (Infections and infestations) | 1 (1) | 1 (1)
Brain herniation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Chest injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Patella fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cardiac output decreased (Investigations) | 0 (0) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperlactacidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3)
Hypervolaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Iron deficiency (Metabolism and nutrition disorders) | 1 (2) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (3) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (3) | 0 (0)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Device breakage (Product Issues) | 0 (0) | 1 (1)
Device dislocation (Product Issues) | 2 (2) | 0 (0)
Device malfunction (Product Issues) | 0 (0) | 2 (2)
Device occlusion (Product Issues) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 2 (2)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 22 (27)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 6 (6)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Therapy change (Surgical and medical procedures) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Artery dissection (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)
Reperfusion injury (Vascular disorders) | 0 (0) | 1 (1)
Shock (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sotatercept (N=86) | Placebo (N=86)
Anaemia (Blood and lymphatic system disorders) | 8 (9) | 6 (6)
Thrombocytopenia (Blood and lymphatic system disorders) | 10 (13) | 7 (8)
Atrial fibrillation (Cardiac disorders) | 5 (6) | 2 (2)
Palpitations (Cardiac disorders) | 8 (9) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 6 (6) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 5 (6)
Diarrhoea (Gastrointestinal disorders) | 19 (23) | 15 (16)
Gingival bleeding (Gastrointestinal disorders) | 9 (10) | 2 (2)
Nausea (Gastrointestinal disorders) | 16 (20) | 13 (16)
Vomiting (Gastrointestinal disorders) | 11 (12) | 4 (5)
Fatigue (General disorders) | 11 (11) | 14 (16)
Influenza like illness (General disorders) | 6 (10) | 2 (3)
Oedema peripheral (General disorders) | 11 (14) | 17 (22)
Pyrexia (General disorders) | 6 (6) | 4 (4)
COVID-19 (Infections and infestations) | 12 (14) | 13 (14)
Nasopharyngitis (Infections and infestations) | 9 (11) | 11 (11)
Respiratory tract infection (Infections and infestations) | 2 (2) | 5 (5)
Urinary tract infection (Infections and infestations) | 7 (11) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 5 (5) | 3 (3)
Haemoglobin increased (Investigations) | 8 (14) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 5 (5)
Hypokalaemia (Metabolism and nutrition disorders) | 14 (15) | 12 (15)
Iron deficiency (Metabolism and nutrition disorders) | 7 (11) | 6 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (9) | 4 (7)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (3) | 5 (7)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 5 (5)
Dizziness (Nervous system disorders) | 8 (9) | 8 (9)
Headache (Nervous system disorders) | 20 (23) | 20 (24)
Insomnia (Psychiatric disorders) | 5 (5) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 6 (8)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 (12) | 17 (23)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 38 (54) | 6 (6)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5)
Erythema (Skin and subcutaneous tissue disorders) | 5 (5) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (8) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 5 (8) | 1 (1)
Telangiectasia (Skin and subcutaneous tissue disorders) | 22 (28) | 3 (5)
Hypotension (Vascular disorders) | 11 (11) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication or disclosure of study results will be permitted except as specified in a separate, written agreement between the Sponsor and the investigator. The Sponsor will comply with the requirements for publication of study results. In accordance with standard editorial and ethical practice, the Sponsor will generally support publication.

DOCUMENTS (2):
  • Study Protocol (2024-04-23): https://cdn.clinicaltrials.gov/large-docs/08/NCT04896008/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-16): https://cdn.clinicaltrials.gov/large-docs/08/NCT04896008/SAP_001.pdf